CLINICAL TRIAL: NCT04821726
Title: Evaluation of the Safety and Efficacy of Drug Eluting Balloon Catheter for the Treatment of Patients With Symptomatic Intracranial Atherosclerosis Stenosis
Brief Title: DEB for Symptomatic Intracranial Atherosclerosis Stenosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yinyi(Liaoning) Biotech Co., Ltd. (Industry)
Collaborators: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LNYY2020001
Record Dates: First submitted 2021-03-14; First posted 2021-03-29 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Cerebral Ischemia; Cerebral Atherosclerosis
MeSH Terms: conditions — Brain Ischemia; Intracranial Arteriosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Drug eluting balloon (Vmoky) (Experimental): A paclitaxel eluting balloon produced by Yinyi (Liaoning) Biotech Co., Ltd. Balloon length: 8-40 mm, diameter：1.25-5.00 mm.
  Interventions: Device: Drug eluting balloon (Vmoky)

INTERVENTIONS:
Device: Drug eluting balloon (Vmoky) — Use Vmoky Drug Eluting Balloon to treat patients with symptomatic intracranial atherosclerosis stenosis

SUMMARY:
A prospective, multi-center, single-arm study to evaluate the safety and efficacy of drug eluting balloon catheter for the treatment of patients with symptomatic intracranial atherosclerotic stenosis.

DETAILED DESCRIPTION:
This is a prospective, multi-center, single-arm study to evaluate the safety and efficacy of drug eluting balloon catheter (Vmoky) produced by Yinyi (Liaoning) Biotech Co., Ltd. for the treatment of patients with symptomatic intracranial atherosclerotic stenosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 80 years old；
2. Symptomatic intracranial artery stenosis, the degree of intracranial diseased artery vascular stenosis measured under cerebral angiography between 70~99% (WASID method)；
3. Symptoms are still recurrent after conservative medication (symptoms refer to stroke and transient ischemic episodes of the brain)，or intracranial artery stenosis combined with remote low perfusion performance (rCBF or rCBV abnormalities) in patients.
4. The stenotic vessels are located in the internal carotid artery (intracranial segment), middle cerebral artery, vertebral artery (intracranial segment), basilar artery, distal blood vessels are normal；
5. Only one lesion needed to be treated；
6. The intracranial artery needed to be treated l art mm in diameter；
7. Pre-expansion must be satisfied: forward blood flow TICI 3 level, pre-expanded guide wire retention, observation for 5 minutes, residual stenosis is still ≤50%; without blood limited dissection；
8. Patients have at least 1 porridge plaque risk factor, including past or existing hypertension, diabetes, hyperlipidemia, smoking;
9. mRS≤3 points；
10. Patients or their guardians are able to understand the purpose of the trial, voluntarily participate in and sign a written informed consent form, and receive follow-up visits from patients.

Exclusion Criteria:

1. Target lesion is in-stent restenosis；
2. Exist lesion stenosis more than 50% out of the target vessel；
3. Intracranial haemorrhage occurred within 3 months (substantial cerebral hemorrhage, large amount of subcranial hemorrhage, subdural/external bleeding)；
4. Acute ischemic stroke has occurred in the last two weeks；
5. Stenosis caused by non-atherosclerosis: e.g. arterial mezzanine, moya-moya disease, vasculitis, radioactive vascular disease or fibrous muscle dysplasia;
6. Severe calcified, angulate and Mori type C lesions, as well as congenital development of thin blood vessels and fenestration；
7. Combine intracranial tumors, aneurysms, or intracranial venous malformations；
8. There are risk factors that can lead to cardiogenic embolism: fibrillation, left-ventricle thrombosis, mycardial infarction within 6 weeks, etc；
9. Uncontrollable hypertension by medication (Systolic pressure≥ystolic pres diastolic blood pressure≥pressurec；
10. Severe combined or unstable conditions, such as severe heart failure, lung failure or kidney failure (serum creatinine>3.0mg/dL (264 μmol/L) or renal cyspheric filtration rate (GFR) <30ml/min), severe liver insequencies, malignant tumors;
11. A history of gastrointestinal haemorrhage or haemorrhagic disease (e.g. idiopathic platelet reduction cyanosis, etc.) or a history of bleeding tendencies within 6 months prior to the signing of the informed consent；
12. Hemoglobin is below 90g/L, plateplates<90×109/L；
13. The International Standardized Rate (INR) >1.5, with unreal corrective bleeding factors；
14. Can not carry out antiplatelet/anticoagulant treatment, with anaesthetic and contrast agent contraindication;
15. The angiography shows that the vascular path is curly, and the device is difficult to reach the target position or to withdraw；
16. Patients known to be allergic to heparin, paclitaxel, contrast, aspirin and clopidogrel, anesthetics;
17. Life expectancy is less than 1 year；
18. Participants in other drug or device clinical trials that have not been completed；
19. A pregnant or lactating woman, or a person planning to become pregnant within one year；
20. Other conditions that the researchers consider patients are not suitable.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Restenosis | 6 months (+60 days)
  Restenosis was defined as greater than 50% stenosis within or immediately adjacent (within 5 mm) to the implanted balloon(s) or stent(s) and greater than 20% absolute luminal loss.

SECONDARY OUTCOMES:
Angiographic success rate | immediately after procedure
  TICI 3 blood flow, residual stenosis no more than 50% after 5 minutes and no flow-limited dissection
The success rate of device | immediately after procedure
  device successfully cross the lesion and inflate, post-procedural residual stenosis no more than 50%, no use of bail-out stent
The success rate of procedure | In-hospital (Maximum 7 days after procedure)
  Base on the device success, there is no stroke or death in-hospital
Target lesion stenosis | 6 months (+60 days) and 12 months (±60 days)
  Calculate the stenosis degree with Quantitative Coronary Angiography (QCA) method
Restenosis | 12 months (±60 days)
  Restenosis was defined as greater than 50% stenosis within or immediately adjacent (within 5 mm) to the implanted balloon(s) or stent(s) and greater than 20% absolute luminal loss.
Stroke events | 30 days (±7 days), 6 months (±60 days) and 12 months (±60 days)
  Number of participants that occur these events
Ischemic stroke and transient ischemic attack (TIA) in the area of the responsible blood vessels | 30 days (±7 days), 6 months (±60 days) and 12 months (±60 days)
  Number of participants that occur these events
Ischemic stroke and transient ischemic attack (TIA) out of the area of the responsible blood vessels | 30 days (±7 days), 6 months (±60 days), 12 months (±60 days)
  Number of participants that occur these events
Non-stroke bleeding | 12 months (±60 days)
  Number of participants that occur this event
Mortality | 30 days (±7 days), 6 months (±60 days) and 12 months (±60 days)
  Number of participants that occur this event
Serious adverse events and adverse events | 12 months (±60 days)
  Number of participants that occur these events

CONTACTS AND LOCATIONS:
Overall Officials: Tianxiao Li, Principal Investigator — Henan Provincial People's Hospital
Locations (1):
- Henan Provincial People's Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No